CLINICAL TRIAL: NCT04205266
Title: IV Iron vs Oral Iron for Treatment of Anemia in Women With Abnormal Uterine Bleeding
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thomas Jefferson University (Other)
Collaborators: AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Rebecca Mercier, Assistant Professor, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19C.864
Record Dates: First submitted 2019-12-12; First posted 2019-12-19 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Anemia, Iron Deficiency; Heavy Menstrual Bleeding
MeSH Terms: conditions — Anemia, Iron-Deficiency; Menorrhagia | interventions — Ferrosoferric Oxide; ferrous sulfate; Iron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- IV Iron (Experimental): Will receive 2 infusions of 510mg of ferumoxytol, administered over 15 minutes, 3-8 days apart
  Interventions: Drug: Ferumoxytol
- Oral Iron (Active Comparator): Will receive 325mg ferrous sulfate tablets daily for 60 days
  Interventions: Drug: Ferrous Sulfate

INTERVENTIONS:
Drug: Ferumoxytol — IV iron infusion
  Other Names: Feraheme
  Arms: IV Iron
Drug: Ferrous Sulfate — oral iron therapy
  Other Names: oral iron
  Arms: Oral Iron

SUMMARY:
This study investigates whether intravenous (IV) iron [Feraheme (ferumoxytol) injection)] is a better treatment than oral iron pills (ferrous sulfate) for correcting anemia in women who have heavy menstrual bleeding and anemia. Investigators will study whether women's blood counts respond better, respond more quickly, and if women prefer the IV treatment or the oral treatment. Women who have heavy menstrual bleeding and anemia will be randomly assigned to receive treatment with either oral iron pills or IV iron infusions. Investigators will then check whether and how quickly the anemia improves, and survey participants on how satisfied they were with the treatment.

DETAILED DESCRIPTION:
Screening: All potential participants will be screened. Screening may take place via a phone call if possible. Menstrual history will be reviewed to ensure potential participants meet study definition of heavy menstrual bleeding (self-described bothersome heavy periods, or >7 bleeding days per month). If the participant is a current or former patient in the Jefferson system, the electronic medical record (EMR) will be reviewed as part of screening. If records are available in the EMR that allow confirmation of anemia via the criteria below, screening may be considered complete, and the potential participant may move to an enrollment visit. If the potential participant does not have any records available to review to confirm anemia, they will be seen for an in-person screening visit. If patient has had evaluation as described immediately below completed elsewhere, that is not accessible in the Jefferson EMR or Care Everywhere system, participant will be asked to provide those records for review, and will be seen for an in-person screening visit.

Records will be reviewed to determine if patient has a recently documented diagnosis of anemia. Records will be reviewed to determine if there has been an appropriate clinical evaluation of AUB, generally considered a pelvic ultrasound within the last 12 months and possibly endometrial biopsy within the last 12 months. Standard clinical criteria will be applied to consider whether an endometrial biopsy is needed to rule out malignancy or hyperplasia prior to enrollment. An endometrial biopsy within 12 months will be required for all women over age 40 who have >7 bleeding days per month. An endometrial biopsy will be required for women under age 40 who have >7 bleeding days per month who have at least one additional risk factor for endometrial hyperplasia: obesity with BMI>30, use of any hormone therapy other than standard contraceptive formulations, reported history of polycystic ovarian syndrome, family history of gynecologic or colon cancers in a first degree relative.

If patient has known anemia (hgb <11.5 documented within 60 days) and is not on any current corrective iron therapy and has had appropriate clinical evaluation, participant will move to the enrollment phase.

If patient does not meet above criteria, further evaluation will be done to ensure enrollment criteria. Any patient who needs any evaluation that involves a procedure as described below, will undergo informed consent for the study at this time.

This evaluation will be targeted to address what is lacking in screening:

* If patient has no confirmed anemia, or has been on therapy for anemia since the most recent complete blood count (CBC), will have a blood draw for CBC to confirm anemia. If anemia is confirmed and there is no other evaluation needed will move to enrollment.
* If patient has not had an ultrasound within the last 12 months it will be scheduled to be performed in our obstetrics and gynecology ultrasound unit or by a study investigator. When this is complete, if no further evaluation is needed she will move onto the enrollment phase.
* If patient has not had an endometrial biopsy within 12 months to evaluate AUB, and meets criteria for needing this as listed above, an endometrial biopsy will be performed by a study investigator. When these results confirm no concern for malignancy or other condition requiring specialist referral or urgent intervention, participant will move to the enrollment phase.

If any patient is found to have findings on ultrasound or biopsy that are determined by the study PI or the patient's primary provider to concerning for endometrial hyperplasia or any form of uterine malignancy, they will not be offered enrollment in the study and will be referred for appropriate care.

Enrollment and randomization and baseline bloodwork: If a patient meets all screening criteria for the study, and needs no further testing, they may proceed to the enrollment and randomization process at the screening visit. If any further testing is required, or patient declines to proceed with enrollment at that time, she will return for a future visit for enrollment procedures.

Informed consent will be obtained for any participant who has not yet had this (if no additional procedures such as blood draw, ultrasound or biopsy were needed to complete screening). Baseline demographics and medical information will be entered into the study record. Randomization will be done via the use of sequentially-numbered sealed envelopes. A member of the study team who will not be involved in the enrollment process will use an online generator to develop a randomization scheme with randomly permuted blocks of 4, 6 and 8. Randomization cards will be created and placed in opaque envelopes. After consent and creation of enrollment study record, the next sequential envelope will be opened, and participant will be assigned to either IV iron or oral (standard) care group.

In both groups: participant will complete baseline Duke Health Profile Quality of Life scale. (Appendix 1 in protocol) Participant will be issued a menstrual diary (Attachment B) and be instructed on completion.

If participant is in the standard care group: CBC will be drawn for baseline level. (If screening CBC was within 7 days of enrollment, that value may be used for baseline). Oral iron tablets (ferrous sulfate 325mg) will be dispensed; a sixty day supply will be given. The participant will be instructed to take one tablet daily, starting that day. Participant will be instructed to bring pill bottles and remaining pills to future visits.

If participant is in the IV iron group: date will be selected for patient to present to the Jefferson Clinical Research Unit (JCRU) for ferumoxytol injection. If that date is within 7 days of this enrollment visit, baseline CBC will be drawn now. If the date is >7 days from enrollment, baseline CBC will be deferred and it will be drawn on the date of the initiation of ferumoxytol treatment. If the screening CBC is within 7 days of the planned initiation of treatment, that screening CBC may be used as the baseline value.

Treatment visits:

Participants in the oral iron group will not have treatment visits, as they will self-administer iron at home.

Participants in the intervention (ferumoxytol) group will present to the Jefferson Clinical Research Unit (JCRU) for ferumoxytol injection. If needed, a baseline CBC will be drawn at the OB-GYN research unit immediately prior to the patient presenting to the JCRU. Each participant will receive 510mg of ferumoxytol 50mL diluted in 200mL of 0.9% sodium chloride, infused over 15minutes while in a seated position. Injection will be administered by the JCRU clinical/research staff. A member of the research team will be present for data collection. Each participant will be observed for any signs of hypersensitivity for 30 minutes. Each participant will have vital signs checked at 15 minutes and 30 minutes after injection, prior to discharge from the clinic. Any hypersensitivity reaction or adverse event will be documented in the study chart.

Participant will return for a second ferumoxytol injection, following the same protocol, 3-8 days (per participant availability) later.

All follow up visits will take place at the OB-Gyn clinical research office.

Follow-up visit 1: 12-16 days after initiation of treatment. Participant will present to the research clinic site. CBC will be drawn. Participant will hand in menstrual diary and be issued a new one. Participant will complete Duke quality of life scale. Participant will complete a scale indicating current satisfaction with treatment (Appendix 2 in protocol). Participant will complete questionnaire assessing side effects or interval adverse events related to treatment (Appendix 4 in protocol). Participants in the standard care (oral iron) group will self-report compliance with therapy.

Follow-up visit 2: 28-32 days after initiation of treatment Participant will present to the research clinic site. CBC will be drawn. Participant will hand in menstrual diary and be issued a new one. Participant will complete Duke quality of life scale. Participant will complete a scale indicating current satisfaction with treatment. Participant will complete questionnaire assessing side effects or interval adverse events related to treatment. Participants in the standard care (oral iron) group will self-report compliance with therapy.

Follow-up visit 3: 55-65 days after initiation of treatment Participant will present to the research clinic site. CBC will be drawn. Participant will hand in menstrual diary. Participant will complete Duke quality of life scale. Participant will complete a scale indicating overall satisfaction with treatment (Appendix 3 in protocol). Participant will complete questionnaire assessing side effects of interval adverse events related to treatment. Participants in the standard care (oral iron) group will self-report compliance with therapy. Complete pill counts to assess compliance will also be done.

During the trial, participants may continue whatever treatment has been initiated by their primary provider for the condition of AUB. Participants may initiate new treatment of AUB through their provider throughout the course of the study. Data on initial, ongoing, or new treatments initiated will be collected. Participants who undergo surgical AUB treatment (dilation and curettage, endometrial ablation, myomectomy, uterine artery embolization, hysterectomy) will still be followed with the above study protocols for the expected 60-day duration. For participants who are planning possible surgical intervention at the time of study enrollment investigators will query whether correction of anemia was identified by their provider as a reason to delay surgery. Expected time to surgical intervention will be collected, and if surgical intervention happens during the 60-day study period, actual time to surgical intervention will be noted. Details of the surgical procedure, and impact on bleeding will be collected.

Any participant who receives a blood transfusion, or any oral therapy patient who receives an IV iron or similar treatment outside of the study session will be terminated from the study at the time of that procedure, due to the potential to confound the primary study outcome.

Any participant who become pregnant during the study will be terminated from the study at the time that diagnosis is made, as physiologic changes of pregnancy may confound the primary study outcome.

For any patient terminated from the study, data collected to that point will be included in final analysis.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-50.
* Heavy menstrual bleeding, defined as self-report of bothersome periods with subjectively heavy flow or frequency greater than 7 bleeding days per month.
* Anemia with hgb <11.5 g/dL

Exclusion Criteria:

* Suspected/confirmed malignancy
* Severe anemia currently requiring transfusion or emergent operative intervention
* Allergy or contraindication to either study drug
* Known iron overload
* Known sickle cell disease

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2020-02-14 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin | 60 days after initiation of treatment
  Blood draw to check complete blood count
Hemoglobin | 30 days after initiation of treatment
  Blood draw with check complete blood count
Hemoglobin | 14 days after initiation of treatment
  Blood draw with check complete blood count

SECONDARY OUTCOMES:
Participant satisfaction with treatment | 60 days after initiation of treatment
  Satisfaction with treatment, as measured on study-specific survey Higher scores indicate higher satisfaction
Quality of Life Score | 60 days after initiation of treatment
  Quality of life, as measured on the Duke Health Profile. Validated scale measuring physical health, mental health, anxiety, depression, pain, and disability; Minimum scores are 0; maximum score is 100 on each sub-scale Higher score indicates better outcome / status

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No